CLINICAL TRIAL: NCT04976751
Title: Real World Study on the Application of Appropriate Electrophysiological Technology in the Diagnosis and Treatment of Andrology Diseases in Northwest China
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Yuan Jianlin-1, professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002020080
Record Dates: First submitted 2021-06-23; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pelvic Pain; Chronic Prostatitis
Keywords: transcutaneous electric nerve stimulation; andrology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Electrophysiological treatment group (Experimental): Two electrodes covered the two acupoints of Zhongliao and Huiyang, one electrode covered the three acupoints of Zhongji, Guanyuan and Qihai, and two skin paste electrodes covered the three acupoints of Sanyinjiao, and connected the electric stimulation therapy instrument for 30 minutes. The intensity was based on the patient's tolerance. 4 weeks before the course of treatment, the treatment was performed once a day, 3 times a week.In the last 4 weeks, 20 times were performed twice a week.Fluoroquinolones and alpha blockers were administered according to the patient's symptoms.
  Interventions: Drug: Percutaneous electrical nerve stimulation treatment
- Regular treatment group (No Intervention): Fluoroquinolones and alpha blockers were administered according to the patient's symptoms.

INTERVENTIONS:
Drug: Percutaneous electrical nerve stimulation treatment — Using the percutaneous electrical nerve stimulation instrument to different points of the body
  Arms: Electrophysiological treatment group

SUMMARY:
To carry out real world research on the application of electrophysiology and other suitable technologies in the prevention and treatment of male diseases in medical institutions at all levels in Northwest China, and establish a database for the prevention and treatment of male diseases in Northwest China, so as to provide a basis for the formulation of guidelines or consensus on the application of electrophysiology for the prevention and treatment of male diseases in China.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the diagnostic criteria of National Institutes of Health (NIH)Ⅲ type prostatitis;
* NIH-CPSI score > 10;
* The symptoms lasted for more than 3 months and failed to respond to drug treatment for more than 1 month;
* Age ≥18 years old and ≤60 years old agrees and signs the informed consent;
* Those who did not receive other similar treatment regimens during treatment.

Exclusion Criteria:

* All kinds of bacterial infection caused by acute or chronic orchitis or epididymitis, acute or chronic prostatitis, lower urinary tract infection;
* Benign prostatic hyperplasia, prostate cancer, neurogenic bladder, urethral malformation or stricture and severe neurosis;
* For patients with local pain as the main manifestation, attention should be paid to the exclusion of other lesions in the lower abdomen, perineum, lsosacral sites, such as ureteral calculi, bladder calculi, inguinal hernia, pubis, varicocele, epididymitis, rectocolic diseases, lsodorsal myofascitis, etc.;
* Complicated with heart, brain, liver and hematopoietic system and other serious primary diseases, local skin infection or skin lesions in the treatment site;
* People who have metal implants in their bodies cannot cooperate, such as patients with mental illness.
* People who are allergic to the treatment of electrical stimulation or allergic to a variety of drugs.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — ≥18 years old and ≤60 years old
Enrollment: 274 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health-Chronic Prostatitis Symptom Index(NIH-CPSI) | through study completion, an average of 1 year
  Improvement rate = [(score before treatment - score at the end of treatment)/score before treatment] ×100% The improvement rate ≥75% was considered to be significant.The improvement rate < 75% and ≥50% were considered to be better.
  The improvement rate < 50% and ≥25% were considered as average efficacy.The improvement rate < 25% indicates poor efficacy.

SECONDARY OUTCOMES:
international prostate symptom score (IPSS) | through study completion, an average of 1 year
  The score improved significantly from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
To carry out real world research on the application of electrophysiology and other suitable technologies in the prevention and treatment of male diseases in medical institutions at all levels in Northwest China, and establish a database for the prevention and treatment of male diseases in Northwest China, so as to provide a basis for the formulation of guidelines or consensus on the application of electrophysiology for the prevention and treatment of male diseases in China.